CLINICAL TRIAL: NCT07374094
Title: Studies of Treatment Effects, Host-Pathogen Responses, and Therapeutic Mechanisms in Clostridioides Difficile Infection
Brief Title: Clostridioides Difficile: Understanding Responses and Treatment Effects
Acronym: CURE-CDI
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Other Study IDs: CURE-CDI
Record Dates: First submitted 2025-12-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile infection; Recurrent Clostridioides difficile infection; Fecal microbiota transplantation; Gut microbiota; Microbiome engraftment; Dysbiosis; Microbial metabolites; Intestinal barrier; Immune response; Antibiotic treatment; Observational study
MeSH Terms: conditions — Clostridium Infections; Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Fecal samples, nasopharyngeal swabs, urine samples, peripheral blood mononuclear cells, blood plasma, colonic biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibiotic treatment: Participants with Clostridioides difficile infection receiving standard antibiotic treatment as part of routine clinical care.
  Interventions: Other: Antibiotic treatment
- Fecal microbiota transplantation (FMT): Participants with Clostridioides difficile infection receiving fecal microbiota transplantation as part of routine clinical care.
  Interventions: Other: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Other: Antibiotic treatment — Standard antibiotic treatment for Clostridioides difficile infection administered as part of routine clinical care, according to clinical guidelines. Treatment selection and duration are determined by the treating physician.
  Groups: Antibiotic treatment
Other: Fecal microbiota transplantation (FMT) — Fecal microbiota transplantation administered as part of routine clinical care for Clostridioides difficile infection. The route of administration is determined by clinical practice and physician decision.
  Groups: Fecal microbiota transplantation (FMT)

SUMMARY:
The goal of this observational study is to learn how different treatments for Clostridioides difficile infection (CDI) work, and which biological mechanisms are involved in recovery. The study will compare standard antibiotic treatment and fecal microbiota transplantation (FMT).

The main questions it aims to answer are:

* How do antibiotic treatment and FMT affect treatment outcome in CDI?
* How does the gut microbiota change during and after treatment?
* Which microbial and metabolic factors are associated with recovery or treatment failure?
* How does treatment affect the intestinal barrier, immune response, and patient-reported quality of life?

Participants with CDI will receive treatment as part of routine clinical care, either antibiotics or FMT. Researchers will follow participants over time and collect biological samples to study treatment effects.

Participants will:

* Provide stool samples during the acute infection and during follow-up
* Have treatment outcomes assessed at 2 and 8 weeks
* Be followed for up to 5 years to study long-term effects
* Provide blood and urine samples during follow-up
* Provide nasal samples to study potential microbiota changes at distant body sites
* Complete questionnaires on symptoms and health-related quality of life
* In a subgroup, undergo repeated sigmoid biopsies to study intestinal mucosal healing

The results are expected to increase understanding of how FMT and antibiotics lead to recovery in CDI and may support improved and more targeted future treatments.

DETAILED DESCRIPTION:
Clostridioides difficile infection (CDI) is a frequent cause of antibiotic-associated colitis and is characterized by high rates of recurrence and, in some patients, refractory disease. Although fecal microbiota transplantation (FMT) is an effective treatment for recurrent and refractory CDI, the biological mechanisms underlying treatment response, early clinical improvement, long-term effects, and vulnerability to subsequent antibiotic exposure remain incompletely understood.

This is an observational study designed to characterize biological and clinical changes associated with standard antibiotic treatment and FMT in patients with CDI. The study will investigate intestinal microbiota composition, microbial metabolites, mucosal and systemic immune responses, intestinal barrier function, and patient-reported outcomes, and relate these findings to clinical disease course and treatment outcome.

Adult patients with symptomatic, microbiologically verified CDI receiving routine clinical care will be included. Treatment decisions, including the use of antibiotics or FMT, are made by the treating physician according to clinical guidelines and are not influenced by study participation. Participants will be followed longitudinally for up to five years.

Biological samples will be collected during the acute CDI episode and at predefined follow-up time points. Stool samples will be obtained to characterize intestinal microbiota composition and metabolic profiles over time. In participants treated with FMT, stool sampling will be more frequent during the first week after treatment to capture early post-treatment changes. Blood samples will be collected for assessment of systemic immune and inflammatory markers. Urine samples will be collected for analysis of metabolites related to intestinal barrier integrity. Nasopharyngeal swabs will be obtained to explore whether modulation of the intestinal microbiota is associated with changes in microbiota composition and immune responses at distant mucosal sites.

In a subgroup of participants deemed suitable by the responsible clinician, repeated lower colonic biopsies will be obtained using sigmoidoscopy. These samples will be used to assess colonic mucosal healing, mucus barrier function, mucosa-associated microbiota, and local immune responses.

Microbiota analyses will include metagenomic sequencing approaches, and metabolomic analyses will be performed on stool and other biological samples. Immune responses will be assessed using biochemical and cellular assays in blood, mucosal tissue, and relevant sample types. Donor fecal material used for FMT will be analyzed and related to recipient outcomes.

Clinical outcomes will be assessed at 2 and 8 weeks after initiation of the current CDI treatment and during long-term follow-up. Disease severity and treatment outcomes, including treatment response, recurrence, refractory disease, and sustained cure, will be classified according to established clinical guidelines. Participants experiencing treatment failure may re-enter sampling schedules corresponding to subsequent treatment courses.

Patient-reported health-related quality of life will be assessed during acute infection and follow-up using validated generic and disease-specific instruments.

This study aims to provide a detailed characterization of biological and clinical processes associated with FMT and antibiotic treatment in CDI, including early and long-term effects, and to support future optimization of microbiota-based therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Symptomatic, microbiologically verified Clostridioides difficile infection
* Receiving inpatient or outpatient care at Umeå University Hospital
* Able and willing to provide written informed consent
* Willing to participate in protocol-driven follow-up for up to 5 years

Exclusion Criteria:

* Age below 18 years
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with symptomatic, microbiologically verified Clostridioides difficile infection receiving inpatient or outpatient care at Umeå University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sustained cure | At follow-up 8 weeks after initiation of the current CDI treatment.
  Number of participants with sustained cure, defined as resolution of Clostridioides difficile infection symptoms after completion of the current treatment course and no recurrence during the 8-week follow-up period.

SECONDARY OUTCOMES:
Number of participants with CDI recurrence | At follow-up 8 weeks after initiation of the current CDI treatment
  Number of participants with Clostridioides difficile infection recurrence during the 8-week follow-up period, classified according to established clinical guidelines.
Intestinal microbiota diversity | Baseline and longitudinal follow-up up to 5 years
  Changes in intestinal microbiota diversity assessed by metagenomic sequencing of stool samples.
Stool short-chain fatty acid concentrations | Baseline and longitudinal follow-up up to 5 years
  Changes in stool short-chain fatty acid concentrations assessed using metabolomic methods.
Colonic mucus barrier function | Baseline and follow-up assessments up to approximately 8 weeks after initiation of the current CDI treatment
  Changes in colonic mucus barrier function assessed by ex vivo measurements of mucus growth rate and mucus layer integrity in colonic biopsy samples obtained from a subgroup of participants.
Circulating markers of intestinal barrier function | Baseline and longitudinal follow-up up to 5 years
  Changes in circulating biomarkers related to intestinal barrier function measured in peripheral blood.
Health-related quality of life | Baseline and longitudinal follow-up up to 5 years
  Patient-reported health-related quality of life assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) health index value (higher values indicate better quality of life).
Health-related quality of life | Baseline and longitudinal follow-up up to 5 years
  Patient-reported health-related quality of life assessed using the Clostridioides difficile Quality of Life Survey (Cdiff32) total score (range 0-100; higher scores indicate better quality of life).
Number of participants with new Clostridioides difficile infection episodes after subsequent antibiotic exposure | From 8 weeks after initiation of the current CDI treatment and up to 5 years
  Occurrence of new Clostridioides difficile infection episodes following exposure to non-CDI antibiotic treatment during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Rasmuson, MD, PhD, Principal Investigator — Umeå University, Department of Clinical Microbiology and Umeå University Hospital, Department of Infectious Diseases
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the clinical and biological data collected in this observational study.